CLINICAL TRIAL: NCT00220376
Title: Long-Term Open-Label Extension Trial for Subjects Completing the Phase 3 Trial of Fesoterodine (SP584) for the Treatment of Overactive Bladder Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP739
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Overactive Bladder Syndrome

INTERVENTIONS:
Drug: SPM 907

SUMMARY:
This trial will provide long-term data on safety, satisfaction and maintenance on therapy of fesoterodine (SPM 907) in subjects with overactive bladder syndrome.

Subjects completing the 12 week treatment period of SP584 had the opportunity to participate if eligibility was confirmed. They received fesoterodine 8mg with the option to reduce the dose to 4mg during scheduled visits, and to increase again to 8mg, a procedure which can be followed on an annual basis.

The primary variables are long-term safety and tolerability, measured by observation and assessment of adverse events and duration on therapy. Further safety variables include the assessment of laboratory parameters, changes in ECG, physical exams and measurement of residual urine.

Secondary efficacy variables included various parameters derived from micturition diaries and the evaluation of Quality of Life questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Overactive Bladder Syndrome

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Derby, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States